CLINICAL TRIAL: NCT06806553
Title: Comparative Effects of Constraint-Induced Movement Therapy (CIMT) with Motor Relearning Program (MRP) and Bobath Approach to Augment Functional Motor Recovery of Chronic Hemiparetic Arm
Brief Title: Constraint-Induced Movement Therapy (CIMT) with Motor Relearning Program (MRP) and Bobath Approach to Augment Functional Motor Recovery of Chronic Hemiparetic Arm
Acronym: CIMT-MRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Ahad, Clinical Demonstrator, University of Lahore Hospital (ULH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/199/08/24
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Hemiparesis; Hemiparesis After Stroke; Motor Function; Upper Limb Function
Keywords: Constraint-Induced Movement Therapy (CIMT); Motor Relearning Program (MRP); Bobath Therapy; Stroke Rehabilitation; Upper Limb Hemiparesis; Motor Function Recovery
MeSH Terms: conditions — Stroke; Paresis | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: For a study comparing the effects of Constraint-Induced Movement Therapy (CIMT) combined with Motor Relearning Program (MRP) and Bobath therapy on functional motor recovery in patients with chronic hemiparesis.
Who Masked: Outcomes Assessor
Masking Description: Single-blinded assessor was considered to minimize bias in outcome measurements. The assessor was unaware of the intervention group assignment for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Constraint-Induced Movement Therapy (CIMT) with the Motor Relearning Program (MRP) (Experimental): Intensive training sessions focusing on the paretic arm. The unaffected arm is constrained using a mitt or sling to encourage using the affected limb. Emphasis on repetitive practice of functional tasks to enhance motor learning and skill acquisition. MRP Components: Standard physiotherapy sessions emphasizing strength, range of motion, and coordination. Task-specific training and neuromuscular re-education to improve motor function. Therapy sessions are conducted five days a week for six weeks, with additional home exercise programs to reinforce skills.
  Interventions: Behavioral: Constraint-Induced Movement Therapy (CIMT) With Motor Relearning Program (MRP)
- Bobath therapy (Experimental): Bobath therapy is a task-oriented approach focusing on balance, postural control, and the facilitation of normal movement patterns to improve motor skills and independence. It aims to inhibit abnormal muscle tone and promote efficient motor strategies.
  Interventions: Behavioral: Bobath Therapy

INTERVENTIONS:
Behavioral: Constraint-Induced Movement Therapy (CIMT) With Motor Relearning Program (MRP) — Intensive training sessions of 3 hours/day for 6 weeks, focusing on functional tasks with the paretic arm while constraining the unaffected arm using a mitt or sling. Implement a constraint on the non-paretic arm to encourage increased use of the affected arm in daily activities. Use shaping techniques to gradually increase the complexity and difficulty of tasks performed with the affected arm (Rahman, 2016).
  MRP: Standard physiotherapy sessions of 1 hour/day for 6 weeks, including exercises for both affected and unaffected arm. Focus on improving strength, range of motion, and coordination through repetitive task practice, neuromuscular re-education and compensatory strategies (Brkić, 2016; Ghrouz et al., 2023).
  Arms: Constraint-Induced Movement Therapy (CIMT) with the Motor Relearning Program (MRP)
Behavioral: Bobath Therapy — The first step in the Bobath approach is a thorough assessment of the individual's movement patterns, muscle tone, strength, coordination, and functional abilities. This assessment helps in identifying specific impairments and setting goals for treatment. Bobath therapists use specific handling techniques to facilitate normal movement patterns and inhibit abnormal muscle tone. These hands-on techniques aim to promote efficient movement and improve motor control. The Bobath approach emphasizes task-oriented training, where functional activities relevant to the individual's daily life are incorporated into therapy sessions. This helps in improving motor skills in a context that is meaningful to the individual (Grozdek Čovčić et al., 2022; Kuciel et al., 2021).
  Arms: Bobath therapy

SUMMARY:
Hemiparesis is a condition characterized by weakness or the inability to move on one side of the body, making it difficult to perform everyday activities like eating or dressing (Iswatun et al., 2022). It is a common after-effect of stroke that causes weakness on one side of the body, limiting movement and affecting all basic activities such as dressing, eating, and walking. Hemiparesis can also be a sign of a stroke, and the side of the body weakened by hemiparesis could be ipsilateral (the same side as the brain injury) or contralateral (the opposite side of the brain injury) (Obman, 2020).

The symptoms of hemiparesis include: Weakness, Difficulty walking, Loss of balance, Muscle fatigue, Difficulty with coordination, Inability to grasp objects. Additionally, a person with hemiparesis may experience trouble maintaining balance, standing, or walking, as well as a tingling or numbing sensation on the weak side (Brandstaedter & Lindenbaum, 2023). Difficulty grabbing things, moving with precision, and lack of coordination can also be present. Hemiparesis is a one-sided muscle weakness that can affect all or most of the anatomical segments on one side of the body (Dantes et al., 2020).

Constraint-Induced Movement Therapy (MCIMT) with combination of Motor Relearning Program (MRP) has significant effects on stroke rehabilitation. CIMT is considered to achieve its beneficial effects through mechanisms such as overcoming learned nonuse and use-dependent neural plasticity. However, in case of Bobath there in no such evidence. Therefore more studies are needed to evaluate the effects of CIMT with MRP and Bobath only in both acute and chronic post-stroke populations. Therefore, the aim of this research is to focus on rehabilitation of hemiparetic arm. This present study compared the effects of CIMT with MRP versus Bobath to Augment Functional Motor Recovery of Chronic Hemiparetic Arm.

DETAILED DESCRIPTION:
To determine the comparative effects of constraint-induced movement therapy (CIMT) with motor relearning program (MRP) and Bobath therapy to augment functional motor recovery of chronic hemiparetic arm.

Study Design: Randomized Control Trial

Study Setting: The data was collected from the University of Lahore Teaching Hospital and Sehat Medical Complex , Lahore.

Study Duration: 9 months after the approval of synopsis.

Sampling technique: It was purposive sampling technique.

Sample size: The sample size was 56 (28 in each group ) in each group calculated through software

Group A (CIMT +MRP)

Group B (Bobath)

Screening: Patients were screened to meet inclusion criteria. The consent form was taken from patients then patients will be randomly allocated into two groups ( 28 in each group).

Randomization: Patients fulfilling the inclusion criteria were randomly divided into experimental and control groups using the computer software.

Blinding: The study was single-blinded. The assessor was unaware of the treatment given to both groups.

Assessment: Data was collected at baseline, third and then at the end of the six week. Baseline assessments was conducted before the intervention. Post-intervention assessments were conducted immediately after the intervention. Statistical analysis included descriptive statistics, normality test and analysis of variance to compare the outcomes between the two groups.

Treatment Plan:

Both CIMT with MRP and Bobath both groups received 6 weeks of therapy, 5 days per week, for 3 hours/day per session. Each session was divided into phases: warm-up, active intervention, cool-down.Therapists monitored participant progress and adjust difficulty levels as needed. Home exercise programs was provided for daily practice.

Ethical Considerations: This study has received ethical approval from the Institutional Review Board (IRB). Informed consent was obtained from all participants.

Data Analysis: Statistical software was used to analyze the data, with appropriate tests employed based on data normality to compare outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic hemiparesis at least 6 months prior to study enrollment (Lang et al., 2016).
* Chronic hemiparesis affecting one arm only (Lang et al., 2016).
* Age between 50 and 65 years old (Lang et al., 2016).
* Patients experiencing functional limitations in upper limb motor function (Gracies et al., 2019).
* Mini-Mental State Examination (MMSE) score ≥ 24 (Page et al., 2007).
* Patients with mild to moderate spasticity (Jan et al., 2019).
* Able to tolerate and participate actively in the assigned intervention (Gracies et al., 2019)

Exclusion Criteria:

* Recent acute medical/surgical condition unrelated to stroke (Lang et al., 2016).
* Severe cognitive impairment or communication difficulties (Lang et al., 2016)
* Uncontrolled pain or spasticity in the affected arm (Lang et al., 2016).
* History of shoulder instability or major orthopedic surgery in the affected arm (Gracies et al., 2019).

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline, mid-intervention (3 weeks), and post-intervention (6 weeks).
  The Fugl-Meyer Assessment (FMA) is a widely used clinical tool designed to evaluate motor impairment, balance, sensation, and joint functioning in individuals with post-stroke hemiplegia. It consists of various items that assess motor function in the upper and lower extremities, providing a comprehensive measure of motor recovery post-stroke.
Modified Ashworth Scale (MAS) | Baseline, mid-intervention (3 weeks), and post-intervention (6 weeks).
  The Modified Ashworth Scale (MAS) is a 6-point scale used to assess spasticity in patients with lesions to the central nervous system. Scores on the MAS range from 0 to 4, where lower scores represent normal muscle tone and higher scores indicate increased spasticity. The MAS assigns a grade of spasticity based on resistance encountered during passive movement, with a grade of 0 indicating no increase in muscle tone and a grade of 4 representing limb rigidity in flexion or extension.

SECONDARY OUTCOMES:
Pain | Baseline, mid-intervention (3 weeks), and post-intervention (6 weeks).
  The Numeric Pain Rating Scale is a widely utilized tool for assessing pain intensity in adults. It operates on an 11-point scale ranging from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable. Higher scores on this scale signify greater pain intensity, making it a straightforward method for patients to communicate their pain levels to healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Sharif, PhD.PT, Principal Investigator — University of Lahore; Arooj Fatima, Phd.PT, Study Director — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lang CE, Strube MJ, Bland MD, Waddell KJ, Cherry-Allen KM, Nudo RJ, Dromerick AW, Birkenmeier RL. Dose response of task-specific upper limb training in people at least 6 months poststroke: A phase II, single-blind, randomized, controlled trial. Ann Neurol. 2016 Sep;80(3):342-54. doi: 10.1002/ana.24734. Epub 2016 Aug 16. PMID 27447365
- [Background] Jan S, Arsh A, Darain H, Gul S. A randomized control trial comparing the effects of motor relearning programme and mirror therapy for improving upper limb motor functions in stroke patients. J Pak Med Assoc. 2019 Sep;69(9):1242-1245. PMID 31511706
- [Background] Grozdek Covcic G, Jurak I, Telebuh M, Macek Z, Bertic Z, Zura N, Grubisic M, Matic H, Tislar MH, Jakus L. Effects of Bobath treatment and specific mobilizations on gait in stroke patients: A randomized clinical trial. NeuroRehabilitation. 2022;50(4):493-500. doi: 10.3233/NRE-210326. PMID 35311720
- [Background] Gracies JM, Pradines M, Ghedira M, Loche CM, Mardale V, Hennegrave C, Gault-Colas C, Audureau E, Hutin E, Baude M, Bayle N; Neurorestore Study Group. Guided Self-rehabilitation Contract vs conventional therapy in chronic stroke-induced hemiparesis: NEURORESTORE, a multicenter randomized controlled trial. BMC Neurol. 2019 Mar 12;19(1):39. doi: 10.1186/s12883-019-1257-y. PMID 30871480
- [Background] Ghrouz A, Guillen-Sola A, Morgado-Perez A, Munoz-Redondo E, Ramirez-Fuentes C, Curbelo Pena Y, Duarte E. The effect of a motor relearning on balance and postural control in patients after stroke: An open-label randomized controlled trial. Eur Stroke J. 2024 Jun;9(2):303-311. doi: 10.1177/23969873231220218. Epub 2023 Dec 29. PMID 38158722